CLINICAL TRIAL: NCT06233708
Title: Association Between Pre-operative Use of Non-selective Beta-blockers With the Risk of Hepatocellular Carcinoma Recurrence Following Liver Transplantation : a Retrospective Cohort Study
Brief Title: Association Between Pre-op Non-Selective Beta-Blockers and Hepatocellular Carcinoma Recurrence Post-Liver Transplant
Status: Completed | Type: Observational
Sponsor: Asan Medical Center (Other)
Collaborators: Korea Health Industry Development Institute (Other Government)
Responsible Party: Principal Investigator, Jun-Gol Song, Professor, Asan Medical Center
Other Study IDs: 2023-0713
Record Dates: First submitted 2024-01-19; First posted 2024-01-31 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Hepatocellular Carcinoma Recurrent; Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- NSBB group: The NSBB group was defined as those who received NSBBs for at least 30 consecutive days within the 3 months prior to LT.
  Interventions: Drug: Non-Selective Beta-Adrenoreceptor Agonists for Systemic Use
- Control group: Those who did not meet the above criteria were classified as the control group.

INTERVENTIONS:
Drug: Non-Selective Beta-Adrenoreceptor Agonists for Systemic Use — Non-selective blocker including Propranolol, Carvedilol PO was prescribed
  Groups: NSBB group

SUMMARY:
The goal of this observational study is to investigate the effect of non-selective beta-blocker (NSBB) on the recurrence of hepatocellular carcinoma (HCC) following liver transplantation in patients who underwent liver transplantation (LT) for treating hepatocellular carcinoma.

The main question[s] it aims to answer are:

* Is the usage of non-selective beta-blocker associated with decreased recurrence of hepatocellular carcinoma following liver transplantation?
* Is the usage of non-selective beta-blocker associated with all-cause mortality following liver transplantation?

Researchers will compare the NSBB group, including patients who received non-selective beta-blocker therapy for at least 30 consecutive days within 3 months prior to liver transplantation more than 30 days prior, with the control group to to see if non-selective beta-blocker treatment is associated with decreased recurrence of hepatocellular carcinoma following liver transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* Underwent liver transplantation for treating hepatocellular carcinoma
* Between Jan. 2008 - May. 2022

Exclusion Criteria:

* Pediatric patients (Age under 18 years)
* Re-transplantation
* Multi-organ transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent liver transplantation at Asan Medical Center between Jan. 2008 - May 2022. Asan Medical Center is a tertiary, teaching hospital of the University of Ulsan College of Medicine, located in Seoul, South Korea.
Sampling Method: Non-Probability Sample
Enrollment: 2092 (Actual)
Dates: Start 2008-01-01 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Kaplan-Meier survival analysis of HCC recurrence at 5-year follow-up | Baseline and 5-year follow-up
  HCC recurrence, which was diagnosed based on pathological or radiographic evidence of new lesions consistent with HCC, and recurrence-free survival was collected and compared using Kaplan-Meier survival analysis.
Multivariate Cox regression analysis of HCC recurrence at 5-year follow-up | Baseline and 5-year follow-up
  Multivariate Cox regression analysis was performed to identify the risk factors for HCC recurrence.

SECONDARY OUTCOMES:
Kaplan-Meier survival analysis of overall survival at 5-year follow-up | Baseline and 5-year follow-up
  Overall survival was collected and compared using Kaplan-Meier survival analysis.
Multivariate Cox regression analysis of overall survival at 5-year follow-up | Baseline and 5-year follow-up
  Multivariate Cox regression analysis was performed to identify the risk factors for overall mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Jun-Gol Song, MD, PhD, Study Chair — Department of Anesthesiology and Pain Medicine, Asan Medical Center

IPD SHARING:
Plan to Share IPD: No